CLINICAL TRIAL: NCT01173133
Title: Skin Flap Visible Light Spectroscopy (VLS) Oximetry for Monitoring Free-Flap Ischemia During Breast Reconstruction and Recovery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spectros Corporation (Industry)
Collaborators: Mills-Peninsula Medical Center (Unknown); Stanford University (Other)
Responsible Party: Clinical Coordinator, Spectros Corporation
Other Study IDs: FLA-001
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Ischemia
Keywords: Free Flap; Surgery; Ischemia; Outcome; Reconstructive Plastic Surgery; Monitoring
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to understand the relevance of tissue oximetry measures of tissue flaps during surgery and during recovery, and to determine if T-Stat is a reliable and early method of detecting compromised flaps.

DETAILED DESCRIPTION:
The tissue saturation of free flaps will be measured before, during, and after surgery and during recovery.

ELIGIBILITY:
Inclusion Criteria:

* Under surgical breast reconstruction
* Informed consent

Exclusion Criteria:

* Failure to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgical breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Flap Failure and Compromise by Tissue Saturation Values (Efficacy) | 72 hours

SECONDARY OUTCOMES:
Oximetric Diagnosis compared to Clinical Diagnosis, Doppler | 72 hours
Device Safety Measures (safety) | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mills Penisula Hospital, Burlingame, California, United States